CLINICAL TRIAL: NCT06971952
Title: Closing the Tuberculosis Diagnosis Gap in Rural and Malnourished Populations
Brief Title: Tuberculosis in Rural and Malnourished Populations
Acronym: TB-RAMP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Burroughs Wellcome (Industry); The American Society of Tropical Medicine and Hygiene (Other)
Responsible Party: Principal Investigator, Ghassan Ilaiwy, Visiting Assistant Professor Department of Medicine, Division of Infectious Diseases and International Health, University of Virginia
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: HSR230322
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Tuberculosis (TB); Undernutrition
Keywords: Tuberculosis; Active case finding; Undernutrition
MeSH Terms: conditions — Tuberculosis; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facility-based Household Contact Screening (No Intervention): a studied, 12-month lead-in period to prospectively measure facility-based household tuberculosis (TB) screening activities in collaboration with TB Clinic Staff at Haydom Lutheran Hospital. Index people with TB (PWTB) will be consecutively recruited to passively track their TB course and that of their household contacts over a 2-month period
- Conditional Cash Transfer Incentive for Household Contact Screening (Active Comparator): Households with index people with TB (PWTB) will be consecutively recruited and offered a conditional cash transfer once all HHCs complete the facility-based tuberculosis (TB) screening procedures. The participants will be notified of the cash transfer during the consenting process for this phase. They will be informed that if all household contacts complete the recommended TB screening, the cash transfer will be given to the head of household during the home visit at 2 months.
  Interventions: Behavioral: Conditional Cash Transfer Incentive for Household Contact Screening

INTERVENTIONS:
Behavioral: Conditional Cash Transfer Incentive for Household Contact Screening — Households with index people with TB (PWTB) will be consecutively recruited and offered a conditional cash transfer once all HHCs complete the facility-based tuberculosis (TB) screening procedures. The participants will be notified of the cash transfer during the consenting process for this phase. They will be informed that if all household contacts complete the recommended TB screening, the cash transfer will be given to the head of household during the home visit at 2 months.
  Arms: Conditional Cash Transfer Incentive for Household Contact Screening

SUMMARY:
Background: Tuberculosis (TB) remains a large public health threat in Tanzania with an estimated incidence of 195 per 100,000 people in 2022 and 36% of cases going undiagnosed. Nutritional and financial barriers combine to compound the burden of TB in Tanzania and many other high burden countries.

Objectives: In this study, we aim to evaluate the effect and cost-effectiveness of conditional cash transfer added to the current facility-based approach to improve TB screening among household contacts (HHCs) of index people diagnosed with TB disease (PWTB) in rural Tanzania; and characterize the prevalence of undernutrition among HHCs of index PWTB and quantify the effect of undernutrition severity on the progression to active TB disease.

Methods: In this prospective, interventional cohort study we plan to enroll 360 PWTB and their households within 2 months of TB treatment initiation. The duration of the study is 3 years in total: 2-year enrollment period, divided equally between the current standard of care phase and the added conditional cash transfer phase. All participating households will be visited 2 months after enrollment to complete TB screening for all HHCs and perform anthropometric measurements, and then followed a 2-year period to evaluate for incident TB disease among HHCs.

Data analysis: The proportion of households completing TB screening procedures for all HHCs during phase 1 will be compared to that during phase 2 using a chi-square test to evaluate the effect of conditional cash transfer on completion of HHC TB screening. A similar approach will be used to compare proportions of HHCs diagnosed with active TB disease based on nutritional status. We will use regression and Bayesian modeling to quantify the effect of demographic, nutritional and socioeconomic predictors on completion of HHC TB screening and the incidence of TB disease among HHCs to prioritize higher risk subgroup for TB prevention effort.

Impact: Successful completion of this proposal will informTB programs in many high burden countries with implementable interventions that can be scaled in rural communities to prioritize TB prevention efforts to the HHCs at the highest risk of developing TB disease

ELIGIBILITY:
Inclusion Criteria:

* Index person/people diagnosed with drug sensitive pulmonary tuberculosis disease (PWTB) and starting TB treatment within 2 months of enrollment, of any age.
* Index PWTB are eligible if they reside within the catchment area of Haydom Lutheran Hospital (HLH), and
* Index PWTB intend to receive TB care at a participating study site.
* Index PWTB (or their parent or guardian if index PWTB are <18 years) and head of household (if different from index PWTB) are able and willing to provide informed consent.

Exclusion Criteria:

* Inability to provide informed consent, or assent when applicable.
* Residing or receiving TB care outside of the catchment area of study sites
* Prior completion of TB screening procedures for all household members.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
TB screening completion for all HHCs before the study-initiated home visit | From enrollment to the time of home visit at 2 months
  TB screening completion for all HHCs before the study-initiated home visit; this is a feasible outcome with significant impact on downstream steps in the TB prevention cascade. Population level statistics related to facility-based TB screening in Manyara region are unpublished. Based on findings from our pilot study, we anticipate conditional cash transfers to achieve >50% completion of TB screening for HHCs compared to <15% at baseline (anticipate improvement of TB screening completion to 15% at baseline compared to the 7% baseline noted prior to our pilot study due to closer follow up)
Quantify the effect of undernutrition severity on the progression to active TB disease | one year
  We anticipate that HHCs with moderate-to-severe undernutrition at baseline will be 60% more likely to develop active TB disease at one year compared to HHCs with appropriate nutritional status. MUAC will have similar performance to other measures of undernutrition in the context of HHC TB screening

SECONDARY OUTCOMES:
The cost-effectiveness of conditional cash transfer added to the current facility-based approach to improve TB screening among HHCs of index PWTB | 20-year time horizon for the cost-effectiveness model
  Formative data on household expenditures and distance to care from our pilot study as well as prospective findings from this study will inform a Markov state transition model of comparative cost-effectiveness that will find a cash-transfer strategy most cost-effective for completion of HHC TB screening

CONTACTS AND LOCATIONS:
Overall Officials: Tania Thomas, MD MPH, Principal Investigator — University of Virginia
Locations (1):
- Haydom Lutheran Hospital, Haydom, Manyara Region, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided